CLINICAL TRIAL: NCT03682718
Title: Vaginal Misoprostol With Intracervical Foley Catheter Versus Vaginal Misoprostol Alone in Induction of Labor at Term Pregnancy
Brief Title: Vaginal Misoprostol With Intracervical Foley Catheter in Induction of Labor
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Abass, Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ase36278
Record Dates: First submitted 2018-09-21; First posted 2018-09-25 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Induction of Labor Affected Fetus / Newborn
Keywords: misoprostol , intracervical Foley catheter , induction of labor , term pregnancy.
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- vaginal misoprostol and intracervical Foley catheter (Experimental): participants will receive misoprostol by the same dose and method. Transcervical Foley catheter (size 16F, with 30ml balloon capacity) will be passed. The catheter will deﬂated, removed and cervix re-assessed if no spontaneous expulsion occurred at 12 hours post- insertion. A new catheter will be passed for another 12 hours, if the Bishop score is less than 8 this will be considered as failure of induction.
  Interventions: Device: Transcervical Foley catheter; Drug: Misoprostol
- vaginal misoprostol (Active Comparator): Misoprostol group; participants will receive 50 μg intravaginal in the posterior vaginal fornix, 25 μg will be given every 4 hours for another two doses, if a satisfactory Bishop score of 8 not reached, patient will take an overnight rest and she will continue induction by the same doses on the next day-provided that there is no ROMs- (this is according to Ain Shams University Protocol) The maximum dose of Misoprostol is 200 μg.
  Oxytocin infusion will not started until 6 hours after the last dose or if there is no adequate contractions obtained.
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Device: Transcervical Foley catheter — combined methods of induction of labor Floey Catheter with misoprstol
  Arms: vaginal misoprostol and intracervical Foley catheter
Drug: Misoprostol — Misoprstol inserted vaginally for induction of labor

SUMMARY:
The aim of present study is to compare the safety and efficacy of vaginal misoprostol versus the combination of vaginal misoprostol and intracervical Foley catheter in induction of labor at term pregnancy.

DETAILED DESCRIPTION:
Cervical status is a good predictor of the likelihood of vaginal delivery when labor is induced. Any induction method is likely to be effective in a woman with a favorable cervix, whereas no method is highly successful when performed in a woman with a cervix that is unfavorable.

The use of a balloon catheter as induction method was first described in 1862 by Trainer. The goal of the catheter was to ripen the cervix through direct mechanical dilatation of the cervical canal and indirectly by increasing endogenous prostaglandin secretion.

Alternatively, Prostaglandins are one of the key players in cervical ripening by a number of different mechanisms.

The aim of present study is to compare the safety and efficacy of vaginal misoprostol versus the combination of vaginal misoprostol and intracervical Foley catheter in induction of labor at term pregnancy.

ELIGIBILITY:
Inclusion Criteria:

Singleton pregnancy Gestational age ≥ 37 weeks (calculated from reliable menstrual dates and/or late first trimester or early second trimester ultrasound) Modified Bishop Score ≥ 5 Valid indication for induction of labor Intact fetal membranes Normal fetal non-stress test cervical dilation less than or equal to 2cm vertex presentation

Exclusion Criteria:

Any contraindication for vaginal delivery (e.g. placenta Previa, accrete ) Any contraindication for induction of labor (e.g. fetal malpersentation, prior uterine surgery) Active labor Antepartum hemorrhage Eclampsia Patients with hemolysis, elevated liver enzymes and low platelets Suspected chorioamnitis Intrauterine growth retardation Multiple gestation Non-reassuring fetal heart rate Continuous contractions more than 3 times in 10 minutes at onset of induction of labor Intrauterine fetal demise Any contraindication for use of misoprostol (e.g. bronchial asthma, drug allergy, History of glaucoma) Any contraindication for use of Foley catheter (already ripped cervix) Rupture of membranes Not consenting

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 120 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
induction delivery time | 48 hours
  time elapsed from start of induction till delivery of the baby

SECONDARY OUTCOMES:
misoprstol dose | 24 hours
  total misoprstol needed in each group
induction active stage time | 24 hours
  time elapsed from induction of labor till reaching 6 cm cervical dialtation
Mode of delivery | 48 hours
  mode od delivery either vaginal or Caesarian Section
Maternal Pyrexia | 48 hours
  fever (Temp > 37.8 ) any time during labor
hypersystole | 48 hours
  one uterine contraction with duration of more than 90 sec.
Tachysystole | 48 hours
  Tachysystole as 5 or more contraction in 10 minutes for two consecutive 10 minutes without FHR abnormalities.

OTHER OUTCOMES:
Neonatal Apgar score | 1 min after delivery
  Neonatal Apgar score
Neonatal Apgar score | 5 min after delivery
  Neonatal Apgar score
Neonatal birth weight | 10 min after delivery
  Neonatal birth weight
neonatal ICU admission | 2 hours after delivery
  Number of neonates in need for ICU admission

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abass, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264